CLINICAL TRIAL: NCT03485404
Title: Effect of Preoperative Vitamin B12 on Post Operative Cognitive Dysfunction in Elderly Patients Undergoing Non-cardiac Surgery: A Multi-Center, Prospective, Randomized, Double-blinded, Controlled Clinical Trial
Brief Title: Preoperative Vitamin B12 and Folic Acid on POCD in Elderly Non-cardiac Surgical Patients
Acronym: B12-POCD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to slow recruiment. Only 40 patients were recruited in four years.
Sponsor: Xijing Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Tang-Du Hospital (Other); Shaanxi Provincial People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Anhui Provincial Hospital (Other Government); Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Lize Xiong, Professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20172057-1
Record Dates: First submitted 2018-03-07; First posted 2018-04-02 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Post Operative Cognitive Dysfunction
Keywords: POCD; vitamin B12; folic acid
MeSH Terms: interventions — mecobalamin; Vitamin B 12; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Central randomization. Groups are marked as A and B with no participants, care provider, investigator and outcome assessors know which group is the drug and which is the placebo. Placebo are made as tablets that mimics the color, shape and size of the drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VB12+FA (Experimental): Patients will receive oral supplementation of 0.5mg methylcobalamin, 3/day and 5 mg folic acid, 1/day for 7 days before non-cardiac surgery.
  Interventions: Drug: methylcobalamin; Drug: Folic Acid; Procedure: non-cardiac surgery; Behavioral: NPB test
- Placebo (Placebo Comparator): Patients with receive oral tablets of placebo for folic acid 1/d and placebo for methylcobalamin 3/d, which look exactly like the interventional drugs as oral supplementation for 7 days before non-cardiac surgery.
  Interventions: Other: Placebo for methylcobalamin; Other: Placebo for folic acid; Procedure: non-cardiac surgery; Behavioral: NPB test
- Non-surgical controls (Other): Age and sex-matched community elderly people are included for two sessions of NPB test evaluation for calculation of POCD incidence as normal control to in Z value calculation of POCd incidence to rule out learning effect.
  Interventions: Behavioral: NPB test

INTERVENTIONS:
Drug: methylcobalamin — methylcobalamin tablets, 0.5mg/tablet, 3 tablets/day.
  Other Names: vitamin B12; VB12
  Arms: VB12+FA
Drug: Folic Acid — folic acid tablets, 5mg/tablet, 1 tablet/day
  Other Names: vitamin B9
  Arms: VB12+FA
Other: Placebo for methylcobalamin — orange tablets that looks exactly like methylcobalamin
  Arms: Placebo
Other: Placebo for folic acid — yellow tablets that looks exactly like folic acid
  Arms: Placebo
Procedure: non-cardiac surgery — patients elective for non-cardiac surgery will undergo scheduled surgery after 7 days of intervention
  Arms: Placebo; VB12+FA
Behavioral: NPB test — participants will accept Mini-Mental State Examination (MMSE), Patient Health Questionnaire (PHQ-9), ADL, and NPB test before intervention, and NPB by discharge or similar time intermittent after the first assessment for non-surgical controls. Also ADL will be tested again through telephone interview at 3 months after discharge.
  Other Names: neuropsychological battery tests; assessment of POCD

SUMMARY:
This study will recruit patients more than 65 years old eligible for non-cardiac surgery. Patients who participate will take either vitamin B12 and folic acid supplementation or placebo for 7 days before surgery. Neuropsychological test battery (NPB) will be tested before intervention and at discharge for determination of Post operative cognitive dysfunction (POCD). Another group of non-surgical elderly participants will also be tested for NPB to account for learning effect in POCD diagnosis. The hypothesis is that preoperative vitamin B12 supplementation will reduce the incidence of POCD in elderly patients undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Vitamin B12 has long been suggested to have neural nutrient effect and widely used in clinical settings for patients with peripheral nerve injury as well as complementary medicine for patients with CNS disorders, including cognitive dysfunction. Evidences showed that, although no significant improvement in cognitive function was observed in healthy elderly after vitamin B12 supplementation, some studies suggested that patients with pre-existing CNS disorder may benefit from Vitamin B12. Post operational cognitive dysfunction (POCD) is severe, and long-lasting complication that affects as high as 53% of patients in high risk surgeries. Age is an independent risk factor for POCD. Researches have shown that serum vitamin B12 level decrease with age, and methylcobalamin (active form of Vitamin B12) content in the frontal cortex of aged patients are lower than that of younger patients. However, there are no report on effect of preemptive supplementation of vitamin B12 on POCD incidence. Therefore, the current research is aimed to explore the preoperative methylcobalamin supplementation (500 mg, 3/day for 7 days before surgery) on incidence of POCD. Folic acid supplementation is a common companion for vitamin B12 treatment in clinical settings because they are in the same methionine cycle, increase of one may result in deficiency of another. So we added 5 mg, 1/day of folic acid with methylcobalamin in the treatment group.

This study will recruit patients more than 65 years old eligible for non-cardiac surgery. Patients who participate will take either vitamin B12 and folic acid supplementation or placebo for 7 days before surgery. Neuropsychological test battery (NPB) will be tested before intervention and at discharge for determination of Post operative cognitive dysfunction (POCD). Another group of non-surgical elderly participants will also be tested for NPB to account for learning effect in POCD diagnosis. The hypothesis is that preoperative vitamin B12 supplementation will reduce the incidence of POCD in elderly patients undergoing non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age equals or over 65
* 2. Scheduled for spinal or joint replacement surgery under general anesthesia，estimated surgery time over 2h.
* 3. Signed written informed consent obtained
* 4. Non-surgical Controls are age and sex - matched community elderly residents.

Exclusion Criteria:

* 1. Disease of the central nervous system that impairs cognitive function, including all kinds of dementia, and depression
* 2. MMSE score < 24
* 3. Received education for less than 5 years
* 4. Currently taking sedative or antidepressant drugs
* 5. Has taken vitamin B12, folic acid or their derivatives (methycobalamin, cobalamin, tetrahydrofolic acid, etc.) within 6 months.
* 6. Has accepted cardiac or neurological surgery within one year.
* 7. Was admitted for other clinical trials within 3 month
* 8. Patients that regularly taking drugs that affect vitamin B absorption, including colchicine, neomycin, salicylate.
* 9. Has severe visual or auditory problems
* 10. Alcohol or drug dependent (alcohol dependent: drank more than 100 mL of Chinese liqueur with alcohol concentration over 40% everyday for the past 3 months).
* 11. Patients that are already admitted for this study can not be admitted the second time, no matter the cause of surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of POCD at discharge or 7 days after operation | at discharge or at 7 days after operation if the patient is not discharged by then
  POCD incidence is defined as two or more test of the neuropsychological battery declined as compared to preoperative baseline.

SECONDARY OUTCOMES:
Activity daily living score | 3 months after operation
  Telephone interview of activity daily living score （14 items， 1-4 points per item, ranging 14-56 points with 56 being the worst-unable to complete any task of everyday living.）
Serum level of vitamin B12, folic acid and homocysteine | Immediately before anesthesia, immediately after surgery and on the morning of postoperative day 1
  Ten ml of venous blood will be collected from patients to test the differences of serum levels of vitamin B12, folic acid and homocysteine to show the effect of preoperative supplementation and surgery stimulation on these parameters.
Serum level of cystatin C and myeloid differentiation protein 2 | Immediately before anesthesia, immediately after surgery and on the morning of postoperative day 1
  Ten ml of venous blood will be collected from patients to test the differences of serum levels of cystatin C and myeloid differentiation protein 2.
Length of hospital stay | Date from hospital admission to hospital discharge. This length is usually around 7-14 days. It may be longer if the patient have one or more complications. The length will be documented at patient discharge, up to 100 weeks.
  to see if our intervention could reduce the total days of patient spent in hospital,
Incidence of in hospital complications | From date of hospital admission to date of hospital discharge after surgery. Usually 7-14 days, assessed up to 100 weeks.
  Overall rate of perioperative major complications including hemorrhage, deep vein thrombosis, cardiovascular complications, respiratory complications, acute kidney injury, infection or second operative needed, during patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (13):
- China (13):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Shanghai 10th People's Hospital, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Forth People's Hospital, Shanghai